CLINICAL TRIAL: NCT02763046
Title: A Randomized, Double-blind, Placebo-controlled Multicenter Study of Secukinumab (AIN457) to Examine the Clinical Efficacy and the NSAID-sparing Effect of Secukinumab Over 16 Weeks in Patients With Ankylosing Spondylitis (ASTRUM)
Brief Title: Study to Examine the Clinical Efficacy and the Nonsteroidal Anti-inflammatory Drug (NSAID)-Sparing Effect of Secukinumab Over 16 Weeks in Patients With Ankylosing Spondylitis
Acronym: ASTRUM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIN457FDE03; 2015-004575-74 (EudraCT Number)
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; NSAID; ASAS; ASAS-NSAID score; Secukinumab
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Secukinumab - delayed NSAID tapering (Experimental): Induction with secukinumab 150 mg s.c. once per week (Week 0, 1, 2, 3 and 4) followed by maintenance with secukinumab 150 mg s.c. every 4 weeks (Week 8, 12, 16 and 20), with intermittent placebo injections at Week 5, 6, 7, 17, 18 and 19 to maintain the blind.
  NSAID tapering allowed from Week 4 (delayed tapering).
  Interventions: Drug: Secukinumab (AIN457) 150 mg s.c.
- Secukinumab - early NSAID tapering (Experimental): Placebo at weeks 0, 1, 2, 3 to maintain the blind; followed by induction with secukinumab 150 mg s.c. once per week (Week 4, 5, 6, 7, 8) and maintenance with secukinumab 150 mg s.c. every 4 weeks (Week 12, 16 and 20), with intermittent placebo injections at Week 17, 18 and 19 to maintain the blind.
  NSAID tapering allowed from Week 4 (early tapering).
  Interventions: Drug: Secukinumab (AIN457) 150 mg s.c.
- Placebo (Placebo Comparator): Placebo s.c. at Week 0, 1, 2, 3, 4, 5, 6, 7, 8 and 12. After the Week 16 assessments of the secondary endpoint had been performed, these patients received weekly doses of secukinumab 150 mg s.c. (Week 16, 17, 18, 19 and 20).
  NSAID tapering allowed from Week 4.
  Interventions: Drug: Placebo - Secukinumab (AIN457) 150 mg s.c.

INTERVENTIONS:
Drug: Secukinumab (AIN457) 150 mg s.c. — Induction: 5 x 150 mg secukinumab s.c. weekly Maintenance: 4 x 150 mg secukinumab s.c. every 4 weeks Delayed NSAID tapering (tapering following 4 weeks of secukinumab treatment).
  Arms: Secukinumab - delayed NSAID tapering
Drug: Secukinumab (AIN457) 150 mg s.c. — Induction: 5 x 150 mg secukinumab s.c. weekly Maintenance: 3 x 150 mg secukinumab s.c. every 4 weeks Early NSAID tapering (tapering at the start of secukinumab treatment).
  Arms: Secukinumab - early NSAID tapering
Drug: Placebo - Secukinumab (AIN457) 150 mg s.c. — Placebo for 15 weeks. From Week 16 on, 5 x 150 mg secukinumab s.c. weekly.
  Arms: Placebo

SUMMARY:
This study assessed the clinical Assessment of SpondyloArthritis international Society (ASAS) 20 response to secukinumab and evaluated to which extent concomitant nonsteroidal anti-inflammatory drug (NSAID) treatment can be reduced in patients treated with secukinumab or placebo following an initial run-in phase of stable NSAID therapy.

DETAILED DESCRIPTION:
This was a phase IV, 20-week, randomized, double-blind, 3-arm, placebo-controlled, parallel-group, multicenter study to examine the clinical response of secukinumab treatment in patients with ankylosing spondylitis as measured by the Assessment of SpondyloArthritis international Society (ASAS) 20 response and the nonsteroidal anti-inflammatory drug (NSAID)-sparing effect. This study evaluated to which extent nonsteroidal anti-inflammatory drug (NSAID) treatment can be reduced between Week 4 and Week 12 in patients randomized to secukinumab 150 mg or placebo following an initial run-in phase of 4 weeks on stable NSAID therapy. Two NSAID tapering approaches were evaluated in this study:

1. an early tapering approach in which NSAID were tapered at the start of secukinumab treatment,
2. a delayed tapering approach in which NSAID were tapered following 4 weeks of secukinumab treatment.

Patients were randomized 1:1:1 to one of the following treatment groups:

* Secukinumab - delayed NSAID tapering: Induction with secukinumab 150 mg s.c. once per week (Week 0, 1, 2, 3 and 4) followed by maintenance with secukinumab 150 mg s.c. every 4 weeks (Week 8, 12, 16 and 20), with intermittent placebo injections at Week 5, 6, 7, 17, 18 and 19 to maintain the blind. NSAID tapering allowed from Week 4 (delayed tapering).
* Secukinumab - early NSAID tapering: Placebo at weeks 0, 1, 2, 3 to maintain the blind; followed by induction with secukinumab 150 mg s.c. once per week (Week 4, 5, 6, 7, 8) and maintenance with secukinumab 150 mg s.c. every 4 weeks (Week 12, 16 and 20), with intermittent placebo injections at Week 17, 18 and 19 to maintain the blind. NSAID tapering allowed from Week 4 (early tapering).
* Placebo: Placebo s.c. at Week 0, 1, 2, 3, 4, 5, 6, 7, 8 and 12. After the Week 16 assessments of the secondary endpoint had been performed, these patients received weekly doses of secukinumab 150 mg s.c. (Week 16, 17, 18, 19 and 20). NSAID tapering allowed from Week 4.

The primary objective of the study was to demonstrate that the efficacy of secukinumab 150 mg subcutaneous (s.c.) injection (with NSAID tapering) is superior to placebo based on the proportion of patients achieving an ASAS20 response at Week 12. To show superiority, both secukinumab treatment arms were pooled and compared against placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of active AS with prior documented radiologic evidence fulfilling the Modified New York criteria for AS
* Active AS assessed by total BASDAI ≥ 4 (0-10) at baseline
* Spinal pain as measured by BASDAI Question 2 ≥ 4 cm on a 0-10 cm numeric rating scale at baseline
* Total back pain as measured by VAS ≥ 40 mm (0-100 mm) at baseline
* Patients should have been on at least 2 different NSAIDs at the highest recommended dose for at least 4 weeks prior to randomization, with an inadequate response or failure to respond, or less if therapy had to be reduced due to intolerance, toxicity or contraindications
* Patients must report regular intake of NSAIDs of at least 50% of the highest recommended dose at Screening.
* Patients with prior TNFα inhibitor therapy must report regular intake of NSAIDs of at least 50% of the highest recommended dose at baseline after the appropriate washout
* Patients are required to be on a stable dose of NSAIDs for at least 2 weeks before randomization
* Patients who have previously been on a TNFα inhibitor will be allowed entry into study after an appropriate wash-out period prior to randomization
* Patients who have been on a TNFα inhibitor (not more than two) must have experienced an inadequate response to previous or current treatment given at an approved dose for at least 3 months prior to randomization or have been intolerant to at least one administration of an anti-TNFα agent.
* Patients taking MTX or sulfasalazine are allowed to continue their medication and must have taken it for at least 3 months and be on a stable dose for at least 4 weeks prior to randomization

Key Exclusion Criteria:

* Chest X-ray or MRI with evidence of ongoing infectious or malignant process.
* Previous exposure to Secukinumab or any other biologic drug directly targeting IL-17 or IL-17 receptor
* Patients previously treated with any biological immunomodulating agents, except those targeting TNFα
* Patients who have taken more than two anti-TNFα agents
* Pregnant or nursing (lactating) women.
* History of ongoing, chronic or recurrent infectious disease or evidence of tuberculosis infection.
* Patients who are intolerant to NSAIDs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- Germany (28):
  - Novartis Investigative Site, Bad Doberan
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Cottbus
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Elmshorn
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Freiberg
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Nienburg
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Püttlingen
  - Novartis Investigative Site, Rendsburg
  - Novartis Investigative Site, Saarbrücken
  - Novartis Investigative Site, Schwerin
  - Novartis Investigative Site, Sendenhorst
  - Novartis Investigative Site, Trier

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Kiltz U, Baraliakos X, Brandt-Jurgens J, Wagner U, Lieb S, Sieder C, Mann C, Braun J. Efficacy and NSAID-sparing effect of secukinumab 150 mg in ankylosing spondylitis: results from phase IV ASTRUM study. Ther Adv Musculoskelet Dis. 2024 Jun 5;16:1759720X241255486. doi: 10.1177/1759720X241255486. eCollection 2024. PMID 38846755
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=716

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 40 investigative sites in Germany.
Pre-assignment Details: Participants were randomized 1:1:1 to one of the following treatment groups: secukinumab 150 mg s.c. with delayed NSAID tapering, secukinumab 150 mg s.c. with early NSAID tapering and placebo.
Period: Overall Study
Arm/Group | Secukinumab - Delayed NSAID Tapering | Secukinumab - Early NSAID Tapering | Placebo
Started | 71 | 70 | 70
Completed | 62 | 65 | 62
Not Completed | 9 | 5 | 8
Not completed — Adverse Event | 5 | 4 | 0
Not completed — Lack of Efficacy | 1 | 1 | 3
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Subject/guardian decision | 2 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab - Delayed NSAID Tapering | Secukinumab - Early NSAID Tapering | Placebo | Total
Number analyzed (Participants) | 71 | 70 | 70 | 211
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.2 (13.36) | 44.1 (11.02) | 45.4 (12.55) | 45.2 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 31 | 89
  Male | 41 | 42 | 39 | 122
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 69 | 67 | 68 | 204
  Black | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 1 | 3
  Other | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Achieved ASAS20 Response in the Pooled Secukinumab Group Compared With the Placebo Group at Week 12
Description: ASAS (Assessment of SpondyloArthritis International Society criteria) 20 response is defined as an improvement from baseline of ≥20% and ≥1 unit on a scale of 0-10 in at least three of the four ASAS main domains and no worsening of ≥20% and ≥1 unit on a scale of 0-10 in the remaining domain. The four main ASAS domains are: Patient's global assessment of disease activity, back pain, function represented by ability to perform specific tasks (from Bath Ankylosing Spondylitis Disease Activity Index [BASDAI]) and inflammation represented by mean duration and severity of morning stiffness.
  Non-responder imputation was applied for missing data.
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS) comprising all subjects from the randomized set to whom study treatment was assigned.
Measure: Count of Participants; unit: Participants
Groups:
- Secukinumab - Pooled: The 2 secukinumab arms (delayed NSAID tapering and early NSAID tapering) pooled.
Arm/Group | Secukinumab - Pooled | Placebo
Number analyzed (Participants) | 141 | 70
Participants | 72 | 31
Statistical Analysis 1: Comparison: Secukinumab - Pooled vs Placebo; Test type: Superiority; p = 0.3512, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.74 to 2.36]

2. Secondary Outcome: Proportion of Patients Who Achieved ASAS20 Response in Each Secukinumab Group (Delayed NSAID Tapering and Early NSAID Tapering) Compared With the Placebo Group
Description: as for outcome 1
Time Frame: Baseline, Week 12, Week 16
Population: FAS comprising all subjects from the randomized set to whom study treatment was assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab - Delayed NSAID Tapering | Secukinumab - Early NSAID Tapering | Placebo
Number analyzed (Participants) | 71 | 70 | 70
Participants
  Week 12 | 37 | 35 | 31
  Week 16 | 40 | 35 | 29
Statistical Analysis 1: Comparison: Secukinumab - Delayed NSAID Tapering vs Placebo; Week 12; Test type: Superiority; p = 0.4010, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.68 to 2.60]
Statistical Analysis 2: Comparison: Secukinumab - Early NSAID Tapering vs Placebo; Week 12; Test type: Superiority; p = 0.4382, Regression, Logistic; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.67 to 2.55]
Statistical Analysis 3: Comparison: Secukinumab - Delayed NSAID Tapering vs Placebo; Week 16; Test type: Superiority; p = 0.0934, Regression, Logistic; Odds Ratio (OR) = 1.78, 95% CI 2-sided [0.91 to 3.50]
Statistical Analysis 4: Comparison: Secukinumab - Early NSAID Tapering vs Placebo; Week 16; Test type: Superiority; p = 0.2619, Regression, Logistic; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.75 to 2.90]

3. Secondary Outcome: Mean Change From Baseline in ASAS-NSAID Score at Week 12
Description: ASAS-NSAID score is used to present the NSAID (nonsteroidal anti-inflammatory drug) intake by considering the type of NSAID, the total dose and the number of days taking NSAID during a period of interest (PI). For the NSAID equivalence scoring system, "no NSAID intake" was set to a score value of 0, and the reference dose of 150 mg/day diclofenac was set to a score value of 100. The Daily diclofenac-equivalent dose score was derived by converting each daily dose of NSAID to a percentage dose equivalent of 150 mg diclofenac. ASAS-NSAID score = (equivalent NSAID score) x (days of intake during PI) x (days per week)/(PI in days).
  A negative change from baseline indicates less NSAID consumption.
Time Frame: Baseline, Week 12
Population: FAS comprising all subjects from the randomized set to whom study treatment was assigned.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Secukinumab - Delayed NSAID Tapering | Secukinumab - Early NSAID Tapering | Placebo | Secukinumab - Pooled
Number analyzed (Participants) | 71 | 70 | 70 | 141
Score on scale | -44.9 (47.32) | -40.3 (71.48) | -31.5 (36.54) | -42.6 (60.53)
Statistical Analysis 1: Comparison: Placebo vs Secukinumab - Pooled; Test type: Superiority; p = 0.0997, Mixed Model for Repeated Measures (MMRM); LS (least square) Mean = -10.29, 95% CI 2-sided [-22.55 to 1.96], Standard Error of Mean 6.25
Statistical Analysis 2: Comparison: Secukinumab - Delayed NSAID Tapering vs Placebo; Test type: Superiority; p = 0.0888, Mixed Model for Repeated Measures (MMRM); LS Mean = -12.30, 95% CI 2-sided [-26.47 to 1.87], Standard Error of Mean 7.23
Statistical Analysis 3: Comparison: Secukinumab - Early NSAID Tapering vs Placebo; Test type: Superiority; p = 0.2484, Mixed Model for Repeated Measures (MMRM); LS Mean = -8.29, 95% CI 2-sided [-22.36 to 5.79], Standard Error of Mean 7.18

4. Secondary Outcome: Mean Change From Baseline in ASAS-NSAID Score in Each Secukinumab Group After 12 Weeks of Exposure (at Week 12 in the Secukinumab-delayed NSAID Tapering Group and at Week 16 in the Secukinumab-early NSAID Tapering Group)
Description: ASAS-NSAID score is used to present the NSAID (nonsteroidal anti-inflammatory drug) intake by considering the type of NSAID, the total dose and the number of days taking NSAID during a period of interest (PI). For the NSAID equivalence scoring system, "no NSAID intake" was set to a score value of 0, and the reference dose of 150 mg/day diclofenac was set to a score value of 100. The Daily diclofenac-equivalent dose score was derived by converting each daily dose of NSAID to a percentage dose equivalent of 150 mg diclofenac. ASAS-NSAID score = (equivalent NSAID score) x (days of intake during PI) x (days per week)/(PI in days).
  A negative change from baseline indicates less NSAID consumption. For this endpoint the analysis was performed after 12 weeks of exposure to secukinumab which was achieved at Week 12 in the secukinumab delayed NSAID tapering group but at Week 16 in the secukinumab early NSAID tapering group.
Time Frame: Baseline, Week 12 (delayed NSAID tapering), Week 16 (early NSAID tapering)
Population: FAS comprising all subjects from the randomized set to whom study treatment was assigned.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Secukinumab - Delayed NSAID Tapering | Secukinumab - Early NSAID Tapering
Number analyzed (Participants) | 71 | 70
Score on scale | -44.9 (47.32) | -42.5 (68.62)
Statistical Analysis 1: Comparison: Secukinumab - Delayed NSAID Tapering vs Secukinumab - Early NSAID Tapering; delayed tapering (W12) vs early tapering (W16); Test type: Superiority; p = 0.7735, Mixed Model for Repeated Measures (MMRM); LS Mean = -2.06, 95% CI 2-sided [-16.11 to 11.98]

5. Secondary Outcome: Mean Change From Baseline in the BASDAI Total Score
Description: The BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) is a participant-reported assessment consisting of 6 questions that relate to 5 major symptoms relevant to ankylosing spondylitis: 1) Fatigue, 2) Spinal pain, 3) Peripheral arthritis, 4) Enthesitis, 5) Intensity, and 6) Duration of morning stiffness. Participants need to score each item with a score from 0 to 10 (captured as a continuous visual analog scale). Total score is obtained from the average of symptom scores ranging 0 (no problem) to 10 (worst problem), with a higher score indicating more severe symptoms.
  A negative change from baseline in the total 0-10 BASDAI score indicates improvement.
Time Frame: Baseline, Week 12, Week 16
Population: FAS comprising all subjects from the randomized set to whom study treatment was assigned.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Secukinumab - Delayed NSAID Tapering | Secukinumab - Early NSAID Tapering | Placebo | Secukinumab - Pooled
Number analyzed (Participants) | 71 | 70 | 70 | 141
Score on scale
  Week 12 | -2.1 (2.16) | -2.0 (2.10) | -1.8 (2.00) | -2.1 (2.12)
  Week 16 | -2.3 (1.90) | -2.0 (1.96) | -1.7 (1.96) | -2.2 (1.93)
Statistical Analysis 1: Comparison: Placebo vs Secukinumab - Pooled; Week 12; Test type: Superiority; p = 0.1926, Mixed Model for Repeated Measures (MMRM); LS Mean = -0.39, 95% CI 2-sided [-0.99 to 0.20], Standard Error of Mean 0.30
Statistical Analysis 2: Comparison: Secukinumab - Delayed NSAID Tapering vs Placebo; Week 12; Test type: Superiority; p = 0.1914, Mixed Model for Repeated Measures (MMRM); LS Mean = -0.46, 95% CI 2-sided [-1.14 to 0.23], Standard Error of Mean 0.35
Statistical Analysis 3: Comparison: Secukinumab - Early NSAID Tapering vs Placebo; Week 12; Test type: Superiority; p = 0.3397, Mixed Model for Repeated Measures (MMRM); LS Mean = -0.33, 95% CI 2-sided [-1.01 to 0.35], Standard Error of Mean 0.34
Statistical Analysis 4: Comparison: Secukinumab - Delayed NSAID Tapering vs Placebo; Week 16; Test type: Superiority; p = 0.0384, Mixed Model for Repeated Measures (MMRM); LS Mean = -0.68, 95% CI 2-sided [-1.33 to -0.04], Standard Error of Mean 0.33
Statistical Analysis 5: Comparison: Secukinumab - Early NSAID Tapering vs Placebo; Week 16; Test type: Superiority; p = 0.2116, Mixed Model for Repeated Measures (MMRM); LS Mean = -0.41, 95% CI 2-sided [-1.05 to 0.23], Standard Error of Mean 0.33

6. Secondary Outcome: Mean Change From Baseline in Health-related Quality of Life as Measured by the Short Form-36 Health Survey (SF-36) Physical Component Summary (PCS) Score
Description: The Short Form-36 Health Survey (SF-36) measures the impact of disease on overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 comprise the physical component of the SF-36 (SF-36 PCS) that is evaluated in this study. Scores on each item 1-4 were summed and averaged (range = 0-100 with higher scores indicating better levels of function and/or better health). A positive change from Baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: FAS comprising all subjects from the randomized set to whom study treatment was assigned.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Secukinumab - Delayed NSAID Tapering | Secukinumab - Early NSAID Tapering | Placebo | Secukinumab - Pooled
Number analyzed (Participants) | 71 | 70 | 70 | 141
Score on scale | 4.8 (7.03) | 6.1 (6.92) | 4.8 (7.43) | 5.5 (6.98)
Statistical Analysis 1: Comparison: Placebo vs Secukinumab - Pooled; Test type: Superiority; p = 0.5384, Mixed Model for Repeated Measures (MMRM); LS Mean = 0.63, 95% CI 2-sided [-1.38 to 2.63], Standard Error of Mean 1.02
Statistical Analysis 2: Comparison: Secukinumab - Delayed NSAID Tapering vs Placebo; Test type: Superiority; p = 0.9251, Mixed Model for Repeated Measures (MMRM); LS Mean = -0.11, 95% CI 2-sided [-2.43 to 2.21], Standard Error of Mean 1.18
Statistical Analysis 3: Comparison: Secukinumab - Early NSAID Tapering vs Placebo; Test type: Superiority; p = 0.2432, Mixed Model for Repeated Measures (MMRM); LS Mean = 1.36, 95% CI 2-sided [-0.93 to 3.66], Standard Error of Mean 1.16

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 4 weeks post-treatment (median duration of 24 weeks).
Description: Any signs or symptoms that occurs from first study drug treatment until 30 days after the last study drug treatment. Adverse events were analyzed by treatment period, i.e., Treatment Period 1 from first study drug administration at baseline through Week 16 (concretely: until the day before the injection of study drug scheduled at visit Week 16) and Treatment Period 2 (from the day of injection at visit Week 16 onwards until study end).
Groups:
- Secukinumab - Delayed NSAID Tapering - Treatment Period 1: Induction with secukinumab 150 mg s.c. once per week (Week 0, 1, 2, 3 and 4) followed by maintenance with secukinumab 150 mg s.c. every 4 weeks (Week 8, 12, 16 and 20), with intermittent placebo injections at Week 5, 6, 7, 17, 18 and 19 to maintain the blind. NSAID tapering allowed from Week 4 (delayed tapering).
  Treatment Period 1: from first study drug administration at baseline through Week 16 (concretely: until the day before the injection of study drug scheduled at visit Week 16). This corresponds to the placebo-controlled period of the study.
- Secukinumab - Early NSAID Tapering - Treatment Period 1: Placebo at weeks 0, 1, 2, 3 to maintain the blind; followed by induction with secukinumab 150 mg s.c. once per week (Week 4, 5, 6, 7, 8) and maintenance with secukinumab 150 mg s.c. every 4 weeks (Week 12, 16 and 20), with intermittent placebo injections at Week 17, 18 and 19 to maintain the blind. NSAID tapering allowed from Week 4 (early tapering).
  Treatment Period 1: from first study drug administration at baseline through Week 16 (concretely: until the day before the injection of study drug scheduled at visit Week 16). This corresponds to the placebo-controlled period of the study.
- Placebo - Treatment Period 1: Placebo s.c. at Week 0, 1, 2, 3, 4, 5, 6, 7, 8 and 12. After the Week 16 assessments of the secondary endpoint had been performed, these patients received weekly doses of secukinumab 150 mg s.c. (Week 16, 17, 18, 19 and 20). NSAID tapering allowed from Week 4.
  Treatment Period 1: from first study drug administration at baseline through Week 16 (concretely: until the day before the injection of study drug scheduled at visit Week 16). This corresponds to the placebo-controlled period of the study.
- Secukinumab - Delayed NSAID Tapering - Treatment Period 2: Induction with secukinumab 150 mg s.c. once per week (Week 0, 1, 2, 3 and 4) followed by maintenance with secukinumab 150 mg s.c. every 4 weeks (Week 8, 12, 16 and 20), with intermittent placebo injections at Week 5, 6, 7, 17, 18 and 19 to maintain the blind. NSAID tapering allowed from Week 4 (delayed tapering).
  Treatment Period 2: from the day of injection at visit Week 16 onwards until study end.
- Secukinumab - Early NSAID Tapering - Treatment Period 2: Placebo at weeks 0, 1, 2, 3 to maintain the blind; followed by induction with secukinumab 150 mg s.c. once per week (Week 4, 5, 6, 7, 8) and maintenance with secukinumab 150 mg s.c. every 4 weeks (Week 12, 16 and 20), with intermittent placebo injections at Week 17, 18 and 19 to maintain the blind. NSAID tapering allowed from Week 4 (early tapering).
  Treatment Period 2: from the day of injection at visit Week 16 onwards until study end.
- Placebo - Treatment Period 2: Placebo s.c. at Week 0, 1, 2, 3, 4, 5, 6, 7, 8 and 12. After the Week 16 assessments of the secondary endpoint had been performed, these patients received weekly doses of secukinumab 150 mg s.c. (Week 16, 17, 18, 19 and 20). NSAID tapering allowed from Week 4.
  Treatment Period 2: from the day of injection at visit Week 16 onwards until study end.
Arm/Group | Secukinumab - Delayed NSAID Tapering - Treatment Period 1 | Secukinumab - Early NSAID Tapering - Treatment Period 1 | Placebo - Treatment Period 1 | Secukinumab - Delayed NSAID Tapering - Treatment Period 2 | Secukinumab - Early NSAID Tapering - Treatment Period 2 | Placebo - Treatment Period 2
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/70 | 0/70 | 0/71 | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 4/71 | 3/70 | 1/70 | 1/71 | 0/70 | 1/70
Other Adverse Events (participants affected / at risk) | 53/71 | 56/70 | 55/70 | 25/71 | 23/70 | 22/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab - Delayed NSAID Tapering - Treatment Period 1 (N=71) | Secukinumab - Early NSAID Tapering - Treatment Period 1 (N=70) | Placebo - Treatment Period 1 (N=70) | Secukinumab - Delayed NSAID Tapering - Treatment Period 2 (N=71) | Secukinumab - Early NSAID Tapering - Treatment Period 2 (N=70) | Placebo - Treatment Period 2 (N=70)
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab - Delayed NSAID Tapering - Treatment Period 1 (N=71) | Secukinumab - Early NSAID Tapering - Treatment Period 1 (N=70) | Placebo - Treatment Period 1 (N=70) | Secukinumab - Delayed NSAID Tapering - Treatment Period 2 (N=71) | Secukinumab - Early NSAID Tapering - Treatment Period 2 (N=70) | Placebo - Treatment Period 2 (N=70)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Monoclonal B-cell lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Monocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 3 | 1 | 0 | 1
Hyperprolactinaemia (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Iritis (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Presbyopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 3 | 1 | 1 | 3
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gingival discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 5 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 2 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site urticaria (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Polyp (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 5 | 2 | 3 | 2 | 1 | 1
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 4 | 3 | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infected bite (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 6 | 13 | 14 | 7 | 5 | 3
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 2 | 2 | 0 | 1 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 4 | 3 | 1 | 1 | 3
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 4 | 0 | 2 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Trichomoniasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 1 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Uterine infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Reactive gastropathy (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Laboratory test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pseudohyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pseudohypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 6 | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 1 | 0
Rheumatic fever (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 12 | 10 | 6 | 4 | 3 | 1
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0
Paresis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Uterine pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 4 | 3 | 4 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT02763046/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT02763046/SAP_001.pdf